CLINICAL TRIAL: NCT02284282
Title: Spinal Bupivacaine/Morphine in Laparoscopic Gastro-intestinal Surgery
Acronym: Salmon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL43488.101.13
Record Dates: First submitted 2014-10-17; First posted 2014-11-06 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2016-12

CONDITIONS: Spinal Bupivacaine/Morphine in Laparoscopic Surgery
Keywords: Spinal Morphine; Laparoscopic GI-surgery; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal injection (Active Comparator): Patients receive spinal injection Bupivacaine/Morphine
  Interventions: Drug: Spinal injection bupivacaine/morphine
- Subcutaneum injection (Placebo Comparator): Placebo subcutaneum injections
  Interventions: Drug: subcutaneum injection lidocaine

INTERVENTIONS:
Drug: Spinal injection bupivacaine/morphine — Spinal injection bupivacaine/morphine in laparoscopic surgery
  Other Names: injection
  Arms: Spinal injection
Drug: subcutaneum injection lidocaine — placebo injection
  Other Names: placebo
  Arms: Subcutaneum injection

SUMMARY:
The objective of this study is to determine if a single spinal shot of morphine can decrease post-operative opioid-use, and thereby decrease opioid side-effects and lead to a quicker recovery after surgery.

DETAILED DESCRIPTION:
We expect that in laparoscopic gastro-intestinal surgery, a single shot spinal with bupicavaine/morphine will result in a better analgesia in hte first 48 hours. Herby the patients will require less systemic opioids, which will decrease the side-effects. Furthermore, we expect the patients to recover quicker and show an earlier mobilisation and a shorter hospital stay.

The objective of this study is to determine if a single spinal shot of morphine can decrease post-operative opioid-use, and thereby decrease opioid side-effects and lead to a quicker recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic Gastro-intestinal surgery

Exclusion Criteria:

* Bariatric surgery, gastric surgery, rectal surgery, kidney failure, aorta-valve stenosis, coagulation disorders, emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Duration of hospital stay | first 48 hours

SECONDARY OUTCOMES:
use of piritramide by PCIA-pump in mg | 48 hours
patient-satisfactory on a 4-point scale | 120 hours/ 5 days
the occurence of side-effects (nausea, pruritus, drowsiness) | 120 hours/ 5 days
time to mobilisation | 120 hours/ 5 days
time to bowel movement | 120 hours/ 5 days
abdominal compliance during laparoscopy in L/mmHg | The compliance will be measured for the duration of the surgery, an expected average of 2 hours.
Difficulty of surgery | The difficulty of surgery will be measured for the duration of the surgery, an expected average of 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: AartJan JW Teunissen, MD, Principal Investigator — Maasstad Hospital; Mark V Koning, MD, Principal Investigator — Maasstad Hospital
Locations (1):
- Maasstad Hospital, Rotterdam, Netherlands

REFERENCES:
- [Background] Koning MV, Teunissen AJW, van der Harst E, Ruijgrok EJ, Stolker RJ. Intrathecal Morphine for Laparoscopic Segmental Colonic Resection as Part of an Enhanced Recovery Protocol: A Randomized Controlled Trial. Reg Anesth Pain Med. 2018 Feb;43(2):166-173. doi: 10.1097/AAP.0000000000000703. PMID 29219935
- See also: Full text — https://journals.lww.com/rapm/Fulltext/2018/02000/Intrathecal_Morphine_for_Laparoscopic_Segmental.8.aspx